CLINICAL TRIAL: NCT04676698
Title: Three Good Things 2020: a Brief Text-based Wellness Intervention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Katherine Gold, Associate Professor of Family Medicine and Associate Professor of Obstetrics and Gynecology, University of Michigan
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: HUM00188399
Record Dates: First submitted 2020-12-15; First posted 2020-12-21 (Actual); Last update posted 2021-12-03 (Actual); Status verified 2021-12

CONDITIONS: Job Related Stress
Keywords: Satisfaction; Depression
MeSH Terms: conditions — Occupational Stress; Personal Satisfaction; Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Three Good Things (Experimental): Three times weekly for three weeks, participants will receive a text-based survey asking them to type or dictate "three good things."
  Interventions: Behavioral: Three Good Things
- Waitlist Control Arm then Three Good Things (Active Comparator): Participants will have surveys in the waiting period for 3 months and then be crossed over to the treatment arm Three Good Things.
  Interventions: Behavioral: Wait list control arm and then Three Good Things

INTERVENTIONS:
Behavioral: Three Good Things — The treatment phase will last 3 weeks. However, participants will complete surveys at baseline and up to 6 months. At the end of the trial the study team will also select a limited number of entries from participants to share some of the "good things" which people listed. These will be edited to ensure writer anonymity and participants will be informed of this plan in the study introduction.
  Arms: Three Good Things
Behavioral: Wait list control arm and then Three Good Things — Surveys will be completed for 3 months prior to treatment and then after treatment.
  Arms: Waitlist Control Arm then Three Good Things

SUMMARY:
This trial will be open to all Michigan Medicine Department of Family Medicine faculty, resident, or staff.

The intervention will consist of asking participants the "3 Good Things" based on positive psychology theory. Participants will be asked to list three things that went well that day and to consider their role in these outcomes. Pre and post surveys will be completed to evaluate this intervention.

At the end of the trial the study team will also select a limited number of entries from participants to share some of the "good things" which people listed. These will be edited to ensure writer anonymity and participants will be informed of this plan in the study introduction.

ELIGIBILITY:
Inclusion Criteria:

* Faculty, resident, or staff in the Michigan Medicine (MM) Department of Family Medicine

Exclusion Criteria:

* Not a member of Family Medicine at MM

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 223 (Actual)
Dates: Start 2021-02-03 (Actual); Primary Completion 2021-08-28 (Actual); Study Completion 2021-08-28 (Actual)

PRIMARY OUTCOMES:
Change in the Positive and Negative Affect Schedule (PANAS-SF) between the intervention and control group | Pre-Treatment (baseline), up to 6 months
  This is a 10 item survey to measure positive and negative affect. Responses include; very slightly or not at all, a little, quite a bit, and extremely. Higher scores of Positive Affect (PA) subscale represent higher positive affect higher scores of Negative affect (NA) subscale represent higher negative affect.

SECONDARY OUTCOMES:
Change in self-reported physical health | Pre-Treatment (baseline), up to 6 months
  This is a 1 question item to assess participants physical health ( 1=Excellent 2=good 3=fair 4=poor).
Change in self-reported mental health | Pre-Treatment (baseline), up to 6 months
  This is a 1 question item to assess participants mental health ( 1=Excellent 2=good 3=fair 4=poor).
Change in Gratitude using the Gratitude Adjective Checklist (GAC) | Pre-Treatment (baseline), up to 6 months
  The GAC is a 3-item self-report measure of state gratitude in which participants select, (1) A little (2) Moderately, Quite a bit (4), and Extremely (5).The total score on GAC ranges from 3 to 15, with higher score indicating greater state gratitude.
Change in depression using the Patient Health Questionnaire 9-item (PHQ-9) score | Pre-Treatment (baseline) to 6 months
  PHQ-9 scores reflect depression severity. Participants will select responses that include 0=not at all, 1=several days, 2=more than half the days, 3=nearly every day. Ranges in scores are from 0-27 (Scores: 0-4 none, 5-9 mild, 10-14 moderate, 15-19 moderately severe, 20-27 severe).
Change in Satisfaction with Life Questionnaire | Pre-Treatment (baseline), up to 6 months
  This is a 5 question questionnaire in which participants select from 7 responses that are given a 1-7 scale from strongly disagree to strongly agree. Scoring ranges from 5-35 where 20 = neutral (the higher the score the more satisfaction).
Change in the Hope Scale | Pre-Treatment (baseline), up to 6 months
  This is a 12 item questionnaire in which participants select from answers that include 1=definitely false 2=mostly false 3=mostly true 4=definitely true.
  Scores range from 12-48 with higher scores indicating greater hope.

CONTACTS AND LOCATIONS:
Overall Officials: Katherine Gold, MD, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No